

Beyond eosinophils: proteomics to identify potential biomarkers of organ damage and response to MEPOLIZUMAB in EGPA

Protocol Number: 14918

Compound Number or Name: BEOMICS study

Brief Title: **Beyond EOsinophils: proteoMICS to identify potential biomarker of organ** damage and response to MEPOLIZUMAB in EGPA

NCT number: n.a.

Date of the document: 12 february 2023